CLINICAL TRIAL: NCT05589064
Title: Evaluation of the Impact of a Dietary and Nutritional Intervention on the Physical, Cognitive, Behavioural and Emotional Symptoms of Patients With Persistent Post-concussive Symptoms
Brief Title: Evaluation of the Impact of a Dietary and Nutritional Intervention on Persistent Post-concussive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de Moncton (Other)
Collaborators: New Brunswick Health Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101616
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Brain Injury Traumatic Mild
Keywords: Dietary intervention; Supplements; Omega-3; Vitamin D; Creatine monohydrate
MeSH Terms: conditions — Brain Concussion | interventions — Cholecalciferol; Creatine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dietary intervention and nutritional supplements (group A) (Experimental): Patients in group A will receive four consultations with a dietitian over eight weeks, in addition to conventional physiotherapy treatments. These patients will receive nutritional counselling and omega-3 (2500mg/day), vitamin D (2000 IU/day) and creatine monohydrate (10mg/day) supplements prescribed by their doctor.
  Interventions: Behavioral: Experimental: Dietetic counseling; Dietary Supplement: Active Comparator: Omega-3, vitamin D3 and creatine monohydrate; Behavioral: Other : Physiotherapy treatment
- Nutritional supplements (group B) (Active Comparator): Patients in group B will be prescribed omega-3 (2500mg/day), vitamin D (2000 IU/day) and creatine monohydrate (10mg/day) supplements and receive physiotherapy treatments over eight weeks.
  Interventions: Dietary Supplement: Active Comparator: Omega-3, vitamin D3 and creatine monohydrate; Behavioral: Other : Physiotherapy treatment
- Physiotherapy treatment (control group) (Other): Patients in the control group will receive physiotherapy treatments over eight weeks.
  Interventions: Behavioral: Other : Physiotherapy treatment

INTERVENTIONS:
Behavioral: Experimental: Dietetic counseling — Patients will receive dietary counselling to increase caloric and nutrient intake, stabilize glycemia, and optimize hydration.
  Arms: Dietary intervention and nutritional supplements (group A)
Dietary Supplement: Active Comparator: Omega-3, vitamin D3 and creatine monohydrate — Patients will be prescribed dietary supplements which will be taken daily for 8 weeks, as per the supplement protocol.
  Arms: Dietary intervention and nutritional supplements (group A); Nutritional supplements (group B)
Behavioral: Other : Physiotherapy treatment — Patients will receive weekly physiotherapy treatment.

SUMMARY:
Concussions affect thousands of Canadians every year. Although the effects are usually temporary, 10-15% of adults experience persistent symptoms likely to last several weeks or even months. It is suggested that nutritional interventions should be considered in concussion management because nutrition can act on several mechanisms of brain injury. However, to date, no study has assessed the impact of dietary interventions on the recovery of people with persistent post-concussive symptoms.

This randomized controlled trial aims to determine the impact of a dietary and nutritional intervention on the physical, cognitive, behavioural and emotional symptoms of patients with persistent post-concussive symptoms in New Brunswick, Canada. Patients will be randomized to one of three groups: 1) dietary treatments and nutritional supplements (experimental group A), 2) nutritional supplements (experimental group B), and 3) physiotherapy treatments (control group). Patients in group A will receive four consultations with a dietitian over eight weeks, in addition to conventional physiotherapy treatments. These patients will receive nutritional counselling and omega-3, vitamin D and creatine supplements. Patients in group B will be prescribed the same supplements as those in group A by their doctor and receive physiotherapy treatments. Finally, patients in the control group will only receive physiotherapy treatments. Patient symptoms will be measured using a questionnaire constructed from tools commonly used in practice. This questionnaire will be completed at the first physiotherapy session and 2, 4 and 8 weeks after the start of the intervention.

DETAILED DESCRIPTION:
Concussions affect thousands of Canadians every year. Although the effects are usually temporary, 10-15% of adults experience persistent symptoms likely to last several weeks or even months. Some studies have explored the impact of pharmaceuticals on treating post-concussive symptoms. Still, these have shown little success, leading the scientific community to consider multidisciplinary approaches to treating and managing concussions. Recently, it has been suggested that nutritional interventions should be considered in concussion management because nutrition can act on several mechanisms of brain injury. Some nutritional supplements have shown beneficial effects on the speed of recovery and the degree of severity of symptoms related to moderate or severe head trauma. Other studies have shown a link between malnutrition and low neurological and cognitive scores. However, to date, no study has assessed the impact of dietary interventions on the recovery of people with persistent post-concussive symptoms.

This randomized controlled trial aims to determine the impact of a dietary and nutritional intervention on the physical, cognitive, behavioural and emotional symptoms of patients with persistent post-concussive symptoms in New Brunswick, Canada. Patients will be randomized to one of three groups: 1) dietary treatments and nutritional supplements (experimental group A), 2) nutritional supplements (experimental group B), and 3) physiotherapy treatments (control group). Patients in group A will receive four consultations with a dietitian over eight weeks, in addition to conventional physiotherapy treatments. These patients will receive nutritional counselling and omega-3, vitamin D and creatine supplements. Patients in group B will be prescribed the same supplements as those in group A by their doctor and receive physiotherapy treatments. Finally, patients in the control group will only receive physiotherapy treatments. The use of three groups will help determine the individual impact of dietetic treatment offered by a dietitian and the use of supplements. Patient symptoms will be measured using a questionnaire constructed from tools commonly used in practice by medical doctors, physiotherapists and dietitians. This questionnaire will be completed at the first physiotherapy session and 2, 4 and 8 weeks after the start of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Must be able to understand English or French
* Have persistent post-concussive symptoms lasting at least 2 weeks but no longer than 6 months

Exclusion Criteria:

* <16 years old
* People who are breastfeeding, pregnant or plan to become pregnant in the next 2 months
* People with neurological disorders (other than concussion) or a history of moderate or severe brain injury
* People in an acute phase of an inflammatory bowel disease
* Any physical condition prohibiting a patient from receiving physiotherapy treatments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in severity of post-concussive symptoms at the end of the intervention | Baseline and Endpoint (Week 8)
  Patients' severity of post-concussive symptoms will be measured using the 5th edition of the Sport Concussion Assessment Tool (SCAT5). This tool assesses the degree of severity of 22 concussion-related symptoms, on a scale of 0 (no symptoms) to 6 (severe). The total number of perceived symptoms is noted by the physiotherapist, and a symptom severity score is calculated (scale from 0 to 132 points).

SECONDARY OUTCOMES:
Change from baseline in balance at the end of the intervention | Baseline and Endpoint (Week 8)
  The physiotherapist will assess patients' balance using the Modified Balance Error Scoring System (mBESS) test. This objective and validated tool is complimentary to the SCAT5 and is scored from 0 to 30 points, where a greater score indicates severe balance impairment.
Change from baseline in vestibular ocular motor at the end of the intervention | Baseline and Endpoint (Week 8)
  The physiotherapist will assess patients' vestibular ocular motor using the Vestibular Ocular Screening (VOMS) test (Mucha et al., 2014). This tool measures five domains, including smooth pursuits, saccades (rapid eye movements), near-point convergence, balance vision reflex and visual motion sensitivity. For each domain, the sum of the symptoms is scored, with a total possible score of 0 (no change) to 200 points (significant changes in symptom severity).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ward Chiasson, PhD, RD, Principal Investigator — Universite de Moncton
Locations (1):
- Universite de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be made available to researchers upon reasonable request made to the principal investigator.

REFERENCES:
- [Background] Ainsley Dean PJ, Arikan G, Opitz B, Sterr A. Potential for use of creatine supplementation following mild traumatic brain injury. Concussion. 2017 Mar 21;2(2):CNC34. doi: 10.2217/cnc-2016-0016. eCollection 2017 Jun. PMID 30202575
- [Background] Aminmansour B, Nikbakht H, Ghorbani A, Rezvani M, Rahmani P, Torkashvand M, Nourian M, Moradi M. Comparison of the administration of progesterone versus progesterone and vitamin D in improvement of outcomes in patients with traumatic brain injury: A randomized clinical trial with placebo group. Adv Biomed Res. 2012;1:58. doi: 10.4103/2277-9175.100176. Epub 2012 Aug 28. PMID 23326789
- [Background] Annweiler C, Milea D, Whitson HE, Cheng CY, Wong TY, Ikram MK, Lamoureux EL, Sabanayagam C. Vitamin D insufficiency and cognitive impairment in Asians: a multi-ethnic population-based study and meta-analysis. J Intern Med. 2016 Sep;280(3):300-11. doi: 10.1111/joim.12491. Epub 2016 Apr 1. PMID 27037788
- [Background] Baltazar GA, Pate AJ, Panigrahi B, LaBoy S, Prosniak R, Mody A, Chendrasekhar A. Malnutrition as measured by albumin and prealbumin on admission is associated with poor outcomes after severe traumatic brain injury. Am Surg. 2015 Feb;81(2):E61-3. No abstract available. PMID 25642858
- [Background] Breck J, Bohr A, Poddar S, McQueen MB, Casault T. Characteristics and Incidence of Concussion Among a US Collegiate Undergraduate Population. JAMA Netw Open. 2019 Dec 2;2(12):e1917626. doi: 10.1001/jamanetworkopen.2019.17626. PMID 31851345
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Cekic M, Cutler SM, VanLandingham JW, Stein DG. Vitamin D deficiency reduces the benefits of progesterone treatment after brain injury in aged rats. Neurobiol Aging. 2011 May;32(5):864-74. doi: 10.1016/j.neurobiolaging.2009.04.017. Epub 2009 May 30. PMID 19482377
- [Background] Cook AM, Peppard A, Magnuson B. Nutrition considerations in traumatic brain injury. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):608-20. doi: 10.1177/0884533608326060. PMID 19033220
- [Background] Curtis L, Epstein P. Nutritional treatment for acute and chronic traumatic brain injury patients. J Neurosurg Sci. 2014 Sep;58(3):151-60. Epub 2014 May 20. PMID 24844176
- [Background] Dolan E, Gualano B, Rawson ES. Beyond muscle: the effects of creatine supplementation on brain creatine, cognitive processing, and traumatic brain injury. Eur J Sport Sci. 2019 Feb;19(1):1-14. doi: 10.1080/17461391.2018.1500644. Epub 2018 Aug 7. PMID 30086660
- [Background] Doroszkiewicz C, Gold D, Green R, Tartaglia MC, Ma J, Tator CH. Anxiety, Depression, and Quality of Life: A Long-Term Follow-Up Study of Patients with Persisting Concussion Symptoms. J Neurotrauma. 2021 Feb 15;38(4):493-505. doi: 10.1089/neu.2020.7313. Epub 2020 Nov 2. PMID 32962513
- [Background] Emanuelson I, Andersson Holmkvist E, Bjorklund R, Stalhammar D. Quality of life and post-concussion symptoms in adults after mild traumatic brain injury: a population-based study in western Sweden. Acta Neurol Scand. 2003 Nov;108(5):332-8. doi: 10.1034/j.1600-0404.2003.00155.x. PMID 14616303
- [Background] Giza CC, Hovda DA. The Neurometabolic Cascade of Concussion. J Athl Train. 2001 Sep;36(3):228-235. PMID 12937489
- [Background] Guskiewicz KM. Assessment of postural stability following sport-related concussion. Curr Sports Med Rep. 2003 Feb;2(1):24-30. doi: 10.1249/00149619-200302000-00006. PMID 12831673
- [Background] Heileson JL, Anzalone AJ, Carbuhn AF, Askow AT, Stone JD, Turner SM, Hillyer LM, Ma DWL, Luedke JA, Jagim AR, Oliver JM. The effect of omega-3 fatty acids on a biomarker of head trauma in NCAA football athletes: a multi-site, non-randomized study. J Int Soc Sports Nutr. 2021 Sep 27;18(1):65. doi: 10.1186/s12970-021-00461-1. PMID 34579748
- [Background] Hou R, Moss-Morris R, Peveler R, Mogg K, Bradley BP, Belli A. When a minor head injury results in enduring symptoms: a prospective investigation of risk factors for postconcussional syndrome after mild traumatic brain injury. J Neurol Neurosurg Psychiatry. 2012 Feb;83(2):217-23. doi: 10.1136/jnnp-2011-300767. Epub 2011 Oct 25. PMID 22028384
- [Background] Institute of Medicine (US) Committee on Nutrition, Trauma, and the Brain; Erdman J, Oria M, Pillsbury L, editors. Nutrition and Traumatic Brain Injury: Improving Acute and Subacute Health Outcomes in Military Personnel. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209314/ PMID 24983072
- [Background] Langer L, Levy C, Bayley M. Increasing Incidence of Concussion: True Epidemic or Better Recognition? J Head Trauma Rehabil. 2020 Jan/Feb;35(1):E60-E66. doi: 10.1097/HTR.0000000000000503. PMID 31246881
- [Background] Lee JM, Jeong SW, Kim MY, Park JB, Kim MS. The Effect of Vitamin D Supplementation in Patients with Acute Traumatic Brain Injury. World Neurosurg. 2019 Jun;126:e1421-e1426. doi: 10.1016/j.wneu.2019.02.244. Epub 2019 Mar 20. PMID 30904798
- [Background] Lewis MD. Concussions, Traumatic Brain Injury, and the Innovative Use of Omega-3s. J Am Coll Nutr. 2016 Jul;35(5):469-75. doi: 10.1080/07315724.2016.1150796. PMID 27454858
- [Background] Lucke-Wold BP, Logsdon AF, Nguyen L, Eltanahay A, Turner RC, Bonasso P, Knotts C, Moeck A, Maroon JC, Bailes JE, Rosen CL. Supplements, nutrition, and alternative therapies for the treatment of traumatic brain injury. Nutr Neurosci. 2018 Feb;21(2):79-91. doi: 10.1080/1028415X.2016.1236174. Epub 2016 Oct 5. PMID 27705610
- [Background] Mah K, Hickling A, Reed N. Perceptions of mild traumatic brain injury in adults: a scoping review. Disabil Rehabil. 2018 Apr;40(8):960-973. doi: 10.1080/09638288.2016.1277402. Epub 2017 Jan 19. PMID 28102739
- [Background] Margulies S, Anderson G, Atif F, Badaut J, Clark R, Empey P, Guseva M, Hoane M, Huh J, Pauly J, Raghupathi R, Scheff S, Stein D, Tang H, Hicks M. Combination Therapies for Traumatic Brain Injury: Retrospective Considerations. J Neurotrauma. 2016 Jan 1;33(1):101-12. doi: 10.1089/neu.2014.3855. Epub 2015 Aug 6. PMID 25970337
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Miller JW, Harvey DJ, Beckett LA, Green R, Farias ST, Reed BR, Olichney JM, Mungas DM, DeCarli C. Vitamin D Status and Rates of Cognitive Decline in a Multiethnic Cohort of Older Adults. JAMA Neurol. 2015 Nov;72(11):1295-303. doi: 10.1001/jamaneurol.2015.2115. PMID 26366714
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780
- [Background] Oliver JM, Jones MT, Kirk KM, Gable DA, Repshas JT, Johnson TA, Andreasson U, Norgren N, Blennow K, Zetterberg H. Effect of Docosahexaenoic Acid on a Biomarker of Head Trauma in American Football. Med Sci Sports Exerc. 2016 Jun;48(6):974-82. doi: 10.1249/MSS.0000000000000875. PMID 26765633
- [Background] Poortmans JR, Francaux M. Adverse effects of creatine supplementation: fact or fiction? Sports Med. 2000 Sep;30(3):155-70. doi: 10.2165/00007256-200030030-00002. PMID 10999421
- [Background] Schneider KJ, Meeuwisse WH, Nettel-Aguirre A, Barlow K, Boyd L, Kang J, Emery CA. Cervicovestibular rehabilitation in sport-related concussion: a randomised controlled trial. Br J Sports Med. 2014 Sep;48(17):1294-8. doi: 10.1136/bjsports-2013-093267. Epub 2014 May 22. PMID 24855132
- [Background] Theadom A, Starkey N, Barker-Collo S, Jones K, Ameratunga S, Feigin V; BIONIC4you Research Group. Population-based cohort study of the impacts of mild traumatic brain injury in adults four years post-injury. PLoS One. 2018 Jan 31;13(1):e0191655. doi: 10.1371/journal.pone.0191655. eCollection 2018. PMID 29385179
- [Background] Vonder Haar C, Peterson TC, Martens KM, Hoane MR. Vitamins and nutrients as primary treatments in experimental brain injury: Clinical implications for nutraceutical therapies. Brain Res. 2016 Jun 1;1640(Pt A):114-129. doi: 10.1016/j.brainres.2015.12.030. Epub 2015 Dec 23. PMID 26723564
- [Background] Wahls T, Rubenstein L, Hall M, Snetselaar L. Assessment of dietary adequacy for important brain micronutrients in patients presenting to a traumatic brain injury clinic for evaluation. Nutr Neurosci. 2014 Nov;17(6):252-9. doi: 10.1179/1476830513Y.0000000088. Epub 2013 Nov 26. PMID 24074905
- [Background] Wu A, Ying Z, Gomez-Pinilla F. The salutary effects of DHA dietary supplementation on cognition, neuroplasticity, and membrane homeostasis after brain trauma. J Neurotrauma. 2011 Oct;28(10):2113-22. doi: 10.1089/neu.2011.1872. Epub 2011 Oct 4. PMID 21851229
- [Background] Wu A, Ying Z, Gomez-Pinilla F. Dietary omega-3 fatty acids normalize BDNF levels, reduce oxidative damage, and counteract learning disability after traumatic brain injury in rats. J Neurotrauma. 2004 Oct;21(10):1457-67. doi: 10.1089/neu.2004.21.1457. PMID 15672635
- [Background] Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms Among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PMID 26954410